CLINICAL TRIAL: NCT05094037
Title: Orthotic Treatment of Diabetic Foot Ulcers: Patient Adherence to Prescribed Wear and Effectiveness of Treatment
Brief Title: Orthotic Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A3781-R
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Counseling

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Treatment group (Experimental): Patients will be given additional counseling
  Interventions: Device: Removable cam walker boot; Other: Counseling
- Control group (Active Comparator): Patients will be given standard of care.
  Interventions: Device: Removable cam walker boot

INTERVENTIONS:
Device: Removable cam walker boot — Standard of care device given to diabetic foot ulcer patients.
Other: Counseling — Additional education, counseling and encouragement of use of the orthosis beyond the current standard of care.
  Arms: Treatment group

SUMMARY:
The United States Department of Veterans Affairs spends an estimated $1.5 billion a year on healthcare for patients with diabetes. The prevalence and complications of diabetes increase with age. Therefore, with the aging of the US and Veteran populations, there is an expectation of increased healthcare costs associated with treating diabetes and the associated complications of this disorder. One common complication is the diabetic foot ulcer. Diabetic foot ulcers are expensive to treat, can take a long time to heal and result in a decrease in patient quality of life. Patients remain susceptible to developing more foot ulcers over time. The goal of this project is to reduce the time it takes to heal a diabetic foot ulcer, increase the time between episodes of ulceration and improve the quality of life for diabetic foot ulcer patients.

ELIGIBILITY:
Inclusion Criteria:

* Veteran patients prescribed an orthotic walking boot for treatment of their diabetic foot ulcer will be eligible to participate in the study.

Exclusion Criteria:

* Veteran patients with amputation proximal to the tarsometatarsal joint, with a Meggitt-Wagner score of 4 or more, with severe infection, with non-ambulatory status or without palpable pedal pulse will be excluded
* All patients will be screened for severe cognitive impairment with the 15 point Brief Interview for Mental Status (BIMS)

  * scores between 12 and 8 will indicate need for extra efforts to support comprehension of instructions, and patients with scores of 7 or less will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Orthosis wear-time | At each clinic visit through study completion, an average of 8 months
  The total time that the orthosis has been worn between clinic visits.
Foot ulcer size | At each clinic visit through study completion, an average of 8 months
  Size of the diabetic foot ulcer.
Foot ulcer healing status | At each clinic visit through study completion, an average of 8 months
  Status of the diabetic foot ulcer.
Number of foot ulcers | At each clinic visit through study completion, an average of 8 months
  The number of diabetic foot ulcers.

CONTACTS AND LOCATIONS:
Overall Officials: Muturi G. Muriuki, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (2):
- United States (2):
  - Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois

IPD SHARING:
Plan to Share IPD: No